CLINICAL TRIAL: NCT03537898
Title: Balanced Solutions and Plasma Electrolytes in the Medical Intensive Care Unit
Brief Title: Balanced Solutions and Plasma Electrolytes
Acronym: BASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Matthew Semler, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 180397
Record Dates: First submitted 2018-05-14; First posted 2018-05-25 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Critical Illness; Acidosis, Metabolic
Keywords: balanced crystalloid; crystalloid; isotonic; acetate; non-acetate; lactated Ringer's; Normosol
MeSH Terms: conditions — Critical Illness; Acidosis | interventions — Ringer's Lactate; normosol R; Plasmalyte A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lactated Ringer's (Active Comparator): Patients in a MICU block randomized to lactated Ringer's will receive lactated Ringer's whenever isotonic intravenous fluid administration is ordered by the treating provider.
  Interventions: Other: Lactated Ringer's
- Normosol (Active Comparator): Patients in a MICU block randomized to Normosol will receive Normosol-R pH 7.4 whenever isotonic intravenous fluid administration is ordered by the treating provider.
  Interventions: Other: Normosol

INTERVENTIONS:
Other: Lactated Ringer's — Lactated Ringer's will be used whenever an isotonic crystalloid is ordered
  Other Names: Ringer's lactate; Non-acetate buffered solution
  Arms: Lactated Ringer's
Other: Normosol — Normosol-R pH 7.4 will be used whenever an isotonic crystalloid is ordered
  Other Names: Normosol-R; Normosol-R pH 7.4; Acetate buffered solution
  Arms: Normosol

SUMMARY:
The administration of intravenous fluids is ubiquitous in the care of the critically ill. Commonly available isotonic crystalloid solutions contain a broad spectrum electrolyte compositions including a range chloride concentrations. Recent prospective, randomized trials have shown improved patient outcomes with the use of balanced crystalloids compared to saline. There have not been large randomized studies comparing acetate buffered balanced crystalloids to non-acetate buffered balanced crystalloids in the critically ill. BASE will be a pilot study for a large, cluster-randomized, multiple-crossover trial enrolling critically ill patients from the Medical ICU at Vanderbilt University from June 2018 until January 2019. The primary endpoint will be plasma bicarbonate concentration between Intensive Care Unit admission and hospital discharge.

DETAILED DESCRIPTION:
BASE is a pilot, cluster-randomized, multiple-crossover trial of lactated Ringer's versus Normosol-R pH 7.4 with regard to plasma bicarbonate concentration between intensive care unit admission and hospital discharge among all patients admitted to the medical intensive care unit. Between June 2018 and January 2019, all patients admitted to the medical intensive care unit at Vanderbilt University Medical Center who are 18 years or older will be enrolled. The study will occur in one-month blocks. The medical intensive care unit (MICU) will be randomized to an initial fluid group (lactated Ringer's or Normosol). The assigned fluid will be used exclusively for all patients receiving isotonic crystalloid for the duration of the month-long block (except in the presence of pre-specified contraindications). The assigned study fluid will switch at the end of each month-long block such that half of hte months are assigned to lactated Ringer's and half of the months are assigned to Normosol-R pH 7.4. It is anticipated that around 2,000 patients will be enrolled from the medical ICU during the study period. The primary outcome analysis will be an intention-to-treat comparison of the primary outcome of bicarbonate concentration (mmol/L) between enrollment and 7 days after enrollment between the lactated Ringer's and Normosol-R groups using generalized estimating equations with a random effect for study period and accounting for repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Medical ICU during the study period (Enrolled patients who are discharged from the hospital are eligible again if they are readmitted to the Medical ICU during the study period)

Exclusion Criteria:

* Age < 18 years old
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2093 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-03-02 (Actual)

PRIMARY OUTCOMES:
Plasma Bicarbonate Concentration | Between ICU admission and Day 7
  The primary outcome is a repeated measures variable of plasma bicarbonate concentration (mmol/L) between ICU admission and 7 days.

SECONDARY OUTCOMES:
Plasma Bicarbonate Concentration < 20 mmol/L | Between ICU admission and Day 7
Lowest Plasma Bicarbonate Concentration | Between ICU admission and Day 7
Plasma Chloride Concentration > 110 mmol/L | Between ICU admission and Day 7
Plasma Chloride Concentration < 100 mmol/L | Between ICU admission and Day 7
Highest Plasma Chloride Concentration | Between ICU admission and Day 7
Change in Plasma Chloride Concentration from Baseline to Peak | Between ICU admission and Day 7
Plasma Sodium Concentration > 145 mmol/L | Between ICU admission and Day 7
Plasma Sodium Concentration < 135 mmol/L | Between ICU admission and Day 7
Plasma Potassium Concentration > 5.5 mmol/L | Between ICU admission and Day 7
Plasma values for Sodium, Potassium, Chloride, Bicarbonate, Blood Urea Nitrogen, Creatinine, Calcium, and Lactate | Between ICU admission and Hospital Discharge or 30 Days
Strong Ion Difference | Between ICU admission and Day 7
  (Sodium + Potassium + Calcium) - (Chloride + Lactate) in mmol/L
Arterial pH | Between ICU admission and Day 7
Arterial Standard Base Excess | Between ICU admission and Day 7
Major Adverse Kidney Events within 30 days | 30 Days after Enrollment Censored at Hospital Discharge
  This composite outcome will be considered present if at least one of the following occur: (1) A patient dies prior to the earlier of hospital discharge or day 30; (2) A patient receives new renal replacement therapy between enrollment and day 30, or (3) A patient has persistent renal dysfunction at the earlier of hospital discharge or day 30 (persistent renal dysfunction is defined as ≥ 200% of creatinine from baseline)
30-Day In-Hospital Mortality | 30 Days after Enrollment Censored at Hospital Discharge
New Renal Replacement Therapy | 30 Days after Enrollment Censored at Hospital Discharge
  The initiation of any renal replacement therapy between enrollment and 30 days censored at hospital discharge in a patient not known to have previously received renal replacement therapy.
Stage II or Higher Acute Kidney Injury | Between ICU admission and Day 7
  A patient will meet this outcome if they meet Kidney Disease Improving Global Outcomes (KDIGO) creatinine criteria for stage II acute kidney injury or higher
Persistent Renal Dysfunction | 30 Days after Enrollment Censored at Hospital Discharge
  Final creatinine value before discharge or 30 days after enrollment ≥ 200% of baseline creatinine.
Total Volume of Blood Product Transfusion | Between ICU admission and Day 7
Dose of Vasopressor | Between ICU admission and Day 7
  Dose of vasopressor (in norepinephrine equivalents, µg/kg/min)
Intensive Care Unit-Free Days | Between ICU admission and Day 28
  Intensive care unit-free days to day 28 (ICU-free days) will be defined as the number of days from the time of the patient's physical transfer out of the ICU until day 28 after enrollment. Patients who die prior to day 28 after enrollment received a value of 0 for ICU-free days. Patients who never transfer out of the ICU prior to day 28 after enrollment will receive a value of 0 for ICU-free days. Patients who transferred out of the ICU, return to the ICU, and are not subsequently transferred out of the ICU again before day 28 after enrollment will receive a value of 0 for ICU-free days. For patients who transfer out of the ICU, are readmitted to the ICU, and subsequently transfer out of the ICU again prior to day 28 after enrollment, ICU-free days will be awarded based on the time of the final transfer out of the ICU prior to day 28 after enrollment.
Vasopressor-Free Days | Between ICU admission and Day 28
  Vasopressor-free days to day 28 will be defined as the number of days from the time of vasopressor cessation until day 28 after enrollment. Patients who die prior to day 28 after enrollment will receive a value of 0 for vasopressor-free days. Patients who never cease to receive vasopressors prior to day 28 after enrollment receive a value of 0 for vasopressor-free days. Patients who achieve vasopressor cessation, return to receiving vasopressors, and do not again achieve vasopressor cessation before day 28 after enrollment receive a value of 0 for vasopressor-free days. For patients who achieve vasopressor cessation, return to receiving vasopressors, and subsequently achieve cessation of vasopressors again prior to day 28 after enrollment, vasopressor-free days will be awarded based on the time of the final cessation of vasopressors prior to day 28 after enrollment. Survivors who never receive vasopressors received 28 vasopressor-free days.
Renal Replacement Therapy-Free Days | Between ICU admission and Day 28
  Renal replacement therapy-free days to day 28 (RRT- free days) will be defined as the number of days from the time of the final RRT treatment until day 28 after enrollment. Patients who die prior to day 28 after enrollment receive a value of 0 for RRT-free days. Patients who continue to receive RRT through day 28 after enrollment receive a value of 0 for RRT-free days. Patients who achieve RRT cessation, return to receiving RRT, and do not again achieve RRT cessation before day 28 after enrollment receive a value of 0 for RRT-free days. For patients who achieve RRT cessation, return to receiving RRT, and subsequently achieve cessation of RRT again prior to day 28 after enrollment, RRT-free days will be awarded based on the time of the final RRT treatment prior to day 28 after enrollment. Survivors who never receive RRT will be awarded 28 RRT-free days.
Ventilator-Free Days | Between ICU admission and Day 28
  Ventilator-free days to day 28 (VFDs) will be defined as the number of days from the time of initiating unassisted breathing (breathing without support of the mechanical ventilator) until day 28 after enrollment. Patients who die prior to day 28 after enrollment will receive a value of 0 for VFDs. Patients who never achieve unassisted breathing prior to day 28 after enrollment will receive a value of 0 for VFDs. Patients who achieve unassisted breathing, returned to assisted breathing, and do not again achieve unassisted breathing before day 28 after enrollment will receive a value of 0 for VFDs. For patients who achieve unassisted breathing, return to assisted breathing, and subsequently achieve unassisted breathing again prior to day 28 after enrollment, VFDs will be awarded based on the time of the final initiation of unassisted breathing prior to day 28 after enrollment. Survivors who never experience assisted breathing will receive 28 VFDs.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Semler, MD, MSc, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finfer S, Liu B, Taylor C, Bellomo R, Billot L, Cook D, Du B, McArthur C, Myburgh J; SAFE TRIPS Investigators. Resuscitation fluid use in critically ill adults: an international cross-sectional study in 391 intensive care units. Crit Care. 2010;14(5):R185. doi: 10.1186/cc9293. Epub 2010 Oct 15. PMID 20950434
- [Background] Semler MW, Self WH, Wanderer JP, Ehrenfeld JM, Wang L, Byrne DW, Stollings JL, Kumar AB, Hughes CG, Hernandez A, Guillamondegui OD, May AK, Weavind L, Casey JD, Siew ED, Shaw AD, Bernard GR, Rice TW; SMART Investigators and the Pragmatic Critical Care Research Group. Balanced Crystalloids versus Saline in Critically Ill Adults. N Engl J Med. 2018 Mar 1;378(9):829-839. doi: 10.1056/NEJMoa1711584. Epub 2018 Feb 27. PMID 29485925
- [Background] Self WH, Semler MW, Wanderer JP, Wang L, Byrne DW, Collins SP, Slovis CM, Lindsell CJ, Ehrenfeld JM, Siew ED, Shaw AD, Bernard GR, Rice TW; SALT-ED Investigators. Balanced Crystalloids versus Saline in Noncritically Ill Adults. N Engl J Med. 2018 Mar 1;378(9):819-828. doi: 10.1056/NEJMoa1711586. Epub 2018 Feb 27. PMID 29485926
- [Background] Weinberg L, Chiam E, Hooper J, Liskaser F, Hawkins AK, Massie D, Ellis A, Tan CO, Story D, Bellomo R. Plasma-Lyte 148 vs. Hartmann's solution for cardiopulmonary bypass pump prime: a prospective double-blind randomized trial. Perfusion. 2018 May;33(4):310-319. doi: 10.1177/0267659117742479. Epub 2017 Nov 16. PMID 29144182
- [Background] Weinberg L, Pearce B, Sullivan R, Siu L, Scurrah N, Tan C, Backstrom M, Nikfarjam M, McNicol L, Story D, Christophi C, Bellomo R. The effects of plasmalyte-148 vs. Hartmann's solution during major liver resection: a multicentre, double-blind, randomized controlled trial. Minerva Anestesiol. 2015 Dec;81(12):1288-97. Epub 2014 Nov 19. PMID 25407026
- [Background] Shin WJ, Kim YK, Bang JY, Cho SK, Han SM, Hwang GS. Lactate and liver function tests after living donor right hepatectomy: a comparison of solutions with and without lactate. Acta Anaesthesiol Scand. 2011 May;55(5):558-64. doi: 10.1111/j.1399-6576.2011.02398.x. Epub 2011 Feb 22. PMID 21342149
- [Background] Hadimioglu N, Saadawy I, Saglam T, Ertug Z, Dinckan A. The effect of different crystalloid solutions on acid-base balance and early kidney function after kidney transplantation. Anesth Analg. 2008 Jul;107(1):264-9. doi: 10.1213/ane.0b013e3181732d64. PMID 18635497
- [Background] Hasman H, Cinar O, Uzun A, Cevik E, Jay L, Comert B. A randomized clinical trial comparing the effect of rapidly infused crystalloids on acid-base status in dehydrated patients in the emergency department. Int J Med Sci. 2012;9(1):59-64. doi: 10.7150/ijms.9.59. Epub 2011 Nov 23. PMID 22211091
- [Derived] Qian ET, Brown RM, Jackson KE, Wang L, Stollings JL, Freundlich RE, Wanderer JP, Siew ED, Bernard GR, Self WH, Casey JD, Rice TW, Semler MW; Pragmatic Critical Care Research Group. Normosol-R vs Lactated Ringers in the Critically Ill: A Randomized Trial. Chest. 2025 Aug;168(2):336-345. doi: 10.1016/j.chest.2025.02.008. Epub 2025 Feb 17. PMID 39971001